CLINICAL TRIAL: NCT02123745
Title: ivWatch Model 400: Device Validation for Infiltrated Tissues
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ivWatch, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IVW400CS-06
Record Dates: First submitted 2014-04-22; First posted 2014-04-28 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2014-06-27 (Estimated); Status verified 2014-05

CONDITIONS: Infiltration of Peripheral IV Therapy
Keywords: infiltration; extravasation; peripheral intravenous therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Infiltrated Tissue (Experimental): The ivWatch Model 400 monitored an IV site during the infiltration of 10 mL of isotonic saline solution. IV sites were placed in the forearm and the dorsal aspect of the hand. The rate of the infiltration ranged between 5 mL/hr to 150 mL/hr.
  Interventions: Device: The ivWatch Model 400

INTERVENTIONS:
Device: The ivWatch Model 400 — The ivWatch Model 400 monitored the site during the course of the infiltration and issued red and/or yellow notifications if an infiltration was detected.

SUMMARY:
A single arm trial consisting of 70 adult volunteers to assess the safety and efficacy of the ivWatch Model 400 when observing infiltrated tissues at common sites for peripheral IV therapy.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Pass health screen by clinician
* 18 years or older

Exclusion Criteria:

* Fail health screen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-02; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ivWatch, LLC, Williamsburg, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Infiltrated Tissue
Started | 71
Completed | 71
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Infiltrated Tissue
Number analyzed (Participants) | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (13.2)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1
  Between 18 and 65 years | 69
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 71
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.2 (6.61)
Skin Pigmentation [Mean (Standard Deviation); unit: units on a scale] — Skin pigmentation was scored from 1 to 3 where 1 represents light skin pigmentation, 2 represents medium skin pigmentation, and 3 represents dark skin pigmentation.
  units on a scale | 1.704 (0.885)

OUTCOME MEASURES:

1. Primary Outcome: Red Notification Sensitivity to Infiltrated Tissues
Description: The ratio of the number of infiltrated IV sites where the ivWatch Model 400 device issued a red notification to the total number of infiltrated IV sites in the study. All infiltrations were limited to 10 mL of isotonic saline solution.
Time Frame: After each participant has been infiltrated, an expected average of 1 hour
Measure: Number (95% Confidence Interval); unit: percentage of infiltrations
Units Other Than Participants: infiltrated IV sites
Arm/Group | Infiltrated Tissue
Number analyzed (Participants) | 70
Number analyzed (infiltrated IV sites) | 140
percentage of infiltrations | 96.4 [91.4 to 98.7]

2. Secondary Outcome: Yellow Notification Sensitivity to Infiltrated Tissues
Description: The ratio of the number of infiltrated IV sites where the ivWatch Model 400 device issued a yellow notification to the total number of infiltrated IV sites in the study. All infiltrations were limited to 10 mL of isotonic saline solution.
Time Frame: After each participant has been infiltrated, an expected average of 1 hour
Measure: Number (95% Confidence Interval); unit: percentage of infiltrations
Units Other Than Participants: infiltrated IV sites
Arm/Group | Infiltrated Tissue
Number analyzed (Participants) | 70
Number analyzed (infiltrated IV sites) | 140
percentage of infiltrations | 99.3 [95.5 to 99.96]

3. Secondary Outcome: Infiltrated Volume When Red Notification Issued
Description: The amount of infiltrated isotonic saline solution when the red notification was issued by the ivWatch Model 400 device.
Time Frame: After each participant has been infiltrated, an expected average of 1 hour
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: infiltrated IV sites
Arm/Group | Infiltrated Tissue
Number analyzed (Participants) | 70
Number analyzed (infiltrated IV sites) | 140
mL | 3.75 (2.13)

4. Secondary Outcome: Infiltrated Volume When Yellow Notification Issued
Description: The amount of infiltrated isotonic saline solution when the yellow notification was issued by the ivWatch Model 400 device.
Time Frame: After each participant has been infiltrated, an expected average of 1 hour
Measure: Mean (Standard Deviation); unit: mL
Units Other Than Participants: infiltrated IV sites
Arm/Group | Infiltrated Tissue
Number analyzed (Participants) | 70
Number analyzed (infiltrated IV sites) | 140
mL | 3.49 (2.04)

5. Secondary Outcome: Significant Skin Irritation or Disruption to Skin Integrity
Description: The number of IV sites that indicated significant skin irritation or disruption to skin integrity assessed at the end of the study.
Time Frame: After each participant has been infiltrated, an expected average of 1 hour
Measure: Number; unit: participants
Arm/Group | Infiltrated Tissue
Number analyzed (Participants) | 70
participants | 0

ADVERSE EVENTS:
Description: Serious and other (non-serious) adverse events were assessed by the clinician performing the study.
Arm/Group | Infiltrated Tissue
Serious Adverse Events (participants affected / at risk) | 0/71
Other Adverse Events (participants affected / at risk) | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes